CLINICAL TRIAL: NCT01040585
Title: Cost Effectiveness Of Linezolid Vs Vancomycin In The Treatment Of Ventilator Acquired Pneumonia In Central America
Brief Title: Cost Effectiveness Of Linezolid In Central America
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5951154
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Ventilator Acquired Pneumonia
Keywords: cost effectiveness; linezolid; ventilator acquired pneumonia; central america
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Central America and the Caribbean: Panama, Costa Rica, Honduras, El Salvador and Nicaragua
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — Treatment for VAP as indication approved and as physician criterium.

SUMMARY:
The therapy with Linezolid (LIN) represents better cost-effectiveness vs. Vancomycin (VAN) for the treatment of nosocomial Pneumonia associate to ventilator (VAP).

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a legally acceptable representative signed and dated informed consent document indicating that him or her has been informed of all pertinent aspects of the study.
* Adult (18 years old or older) men and women with confirm diagnosis of VAP treated on ICU with LIN or VAN; on the selected institutions.

Exclusion Criteria:

* Adult men or women with nosocomial pneumonia not associated to a ventilator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women with VAP.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The rate of resistance Empirical treatment days before specific therapy. Treatment days with Linezolid. Treatment days with Vancomycin. | 4 months
Rate of renal failure. | 4 months
Rate of healing with Linezolid. | 4 months
Rate of healing with Vancomycin. | 4 months

SECONDARY OUTCOMES:
Hospitalization days average with VAN and Linezolid. | 4 months
Variation of prices and values among the different institutions. | 4 months
The average costs of each intervention. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951154&StudyName=Cost%20Effectiveness%20Of%20Linezolid%20In%20Central%20America